CLINICAL TRIAL: NCT00579202
Title: The Gambro Polyflux HD-C4 Small Ease of Use Study
Brief Title: Ease of Use Study for the Gambro Polyflux HD-C4 Small Dialyzer
Status: Completed | Type: Observational
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-0002
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hemodialysis
Keywords: Dialyzer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Gambro HD-C4 Small Dialyzer — Involves the use of FDA 510(k) cleared hemodialyzers and will have no impact on the patient's routine dialysis therapy.

SUMMARY:
The purpose of the study is to study the ease of use of the Polyflux HD-C4 Small dialyzer under conditions of routine clinical use for hemodialysis

DETAILED DESCRIPTION:
Market evaluation protocol.

This ease of use study involves the use of FDA 510(k) cleared hemodialyzers and will have no impact on the patient's routine dialysis therapy. This study is strictly aimed at obtaining feedback from the nursing and technical staff regarding the use of the Polyflux HD-C4 Small dialyzer. The dialysis nursing staff will complete ease of use assessments following routine dialysis therapy.

ELIGIBILITY:
Inclusion Criteria:

* n/a routine dialysis patients

Exclusion Criteria:

* n/a routine dialysis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The dialysis nursing staff will complete ease of use assessments following routine dialysis therapy of adult (≥ 18 years of age) patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
For each dialyzer, the perceived ease of priming. | During priming of each dialyzer

SECONDARY OUTCOMES:
Visual assessment of residual blood in the dialyzer after rinse-back and if dialyzer clotted during treatment. | At the completion of each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rana Irmindra, M.D., Principal Investigator — Advanced Dialysis Center
Locations (1):
- Advanced Dialysis Center, Lanham, Maryland, United States